CLINICAL TRIAL: NCT03539978
Title: Peds SM-THINk (Self-Management Transition to Home INtervention): Nursing Interventions to Improve Discharge Outcomes
Brief Title: Peds SM-THINk: Nursing Interventions to Improve Discharge Outcomes
Acronym: SM-THINk
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Clinical & Translational Science Institute (Unknown); Marquette University (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Stacee Lerret, Associate Professor, Medical College of Wisconsin
Other Study IDs: 1118599
Record Dates: First submitted 2018-04-25; First posted 2018-05-30 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SM-THINk Unit: Two of the three inpatient floors will use the SM-THINk enhanced discharge method. This is part of a clinical practice change and not for research. Parents will complete a questionnaire at the time of the patient's discharge from the hospital.
  Interventions: Other: SM-THINk
- Control Unit: One of the three inpatient floors will use the usual discharge method. Parents will also complete a questionnaire at the time of the patient's discharge from the hospital.

INTERVENTIONS:
Other: SM-THINk — Patients will receive the SM-THINk enhanced discharge method.
  Groups: SM-THINk Unit

SUMMARY:
This study focuses on the delivery of discharge education by clinical nurses to improve parent and family self-management in the home environment. This study tests an discharge method (SM-THINk protocol) designed to improve the quality of care for hospitalized pediatric patients at the time of discharge, enhance the child's and family's experience, and decrease length of stay and health care utilization (ED visit or re-admission). The SM-THINk protocol is an enhancement to the standard clinical practice and will be implemented for all subjects on two Children's Hospital of Wisconsin (CHW) nursing units. This enhancement will require additional training of the nurses prior to implementation of the research project. This research determines the effectiveness of the training enhanced discharge method. The training is independent from the research project and will evaluate effectiveness of this training. For the enhanced discharge method, clinical nurses on the study units will be trained to deliver the Self-Management Transition to Home (SM-THINk protocol), which is based on the family self-management discharge preparation previously developed and tested by the study team.

DETAILED DESCRIPTION:
This quasi-experimental study uses a cluster design with parents from 3 nursing units at the Children's Hospital of Wisconsin. Implementation of the SM-THINk protocol will occur on 2 pediatric inpatient units and a third unit will serve as the usual care control unit. The SM-THINk protocol will be implemented on the two implementation experimental units regardless of this study as a clinical practice change. The nurses will not serve as subjects in this study since they are expected to learn the protocol as part of their everyday jobs.

Plan to enroll 300 patients and one legal guardian per patient (parent or caregiver who has guardianship of the patient). 300 parents of patients per unit (for a total of 900 patients and 900 parents). A high-risk discharge assessment based on Mayo Clinic criteria is used to identify children with complex or chronic conditions. Approximately 120 patients per unit (40%) will have a complex or chronic condition. Parent experience related to quality of discharge teaching and care coordination will be self-reported by parents using established, reliable and valid scales. Child and parent characteristics, length of hospitalization, readmission, and Emergency Department use data will be extracted from electronic medical records.

Nurses on the three units will provide a brief information sheet to families at some point after admission and explain that if the subjects/families have questions that they should call the research team or ask the nurse to contact the research team on their behalf. This information sheet includes a summary of the research purposes and what questions will be asked. When a nurse on the implementation unit is ready to discharge a family who agree to participate, he/she will obtain the iPad, enter the patient code and write down which code corresponds to which patient on a log, perform the enhanced discharge method per clinical practice, then log out of the iPad. He/she will then log into the parent questionnaires (REDCap), enter the patient code, and provide the iPad to the subjects/families. The nurse will indicate that if they would like to participate, they should do so after he/she leaves the room and log out of the iPad when finished. Nurses on the control unit will perform their usual discharge and then obtain the iPad, enter the patient code and write down which code corresponds to which patient on a log. He/she will then log into the parent questionnaires (REDCap), enter the patient code, and provide the iPad to the subjects/families. The nurse will indicate that if they would like to participate, they should do so after he/she leaves the room and log out of the iPad when finished. After approximately 10 minutes the nurse will check to be sure the subject/family has left and if so, will pick up the iPad, ensure the family has logged out, and return the iPad to the storage area. If the subject/family has not left yet, the nurse will check back periodically until they have left. This design will ensure that nursing discharge time is not affected. The research team will pick up the list of patient codes on the next working day. There is a waiver for documentation of informed consent and assent. If the parent and child are interested, participation will serve as implied consent. A HIPAA waiver will be requested by the study team to abstract data from the patient's medical record to look for outcomes over time regarding readmissions and ED visits. Only the following data will be collected from the patient's medical record: the number of hospitalizations in the last 1 year, date of admission/discharge, and the reason for hospitalizations.

All units will ask the parents to complete the parent experience tools at time of discharge using the iPad. Both groups will receive standard post-discharge follow-up care including laboratory and clinic appointments.

The parent's age, insurance information and the child's chronic conditions will all be asked for in the REDCap questionnaires on the iPad. If the iPad is temporarily unavailable for subject/families, paper forms will be provided to them and they will be instructed by the nurses to fill out the forms and seal them in an envelope when they are finished. Nursing staff will provide the sealed envelopes to the research team.

ELIGIBILITY:
A parent/caregiver will be eligible for participation upon meeting the following:

Inclusion Criteria:

1. the parent's/caregiver's child is inpatient on the selected study units
2. the parent/caregiver is English speaking (to date the tools being used have been validated for English participants only)
3. the parent/caregiver is 18 years of age or older
4. the patient is 17 years of age or younger

Exclusion Criteria:

1. presence of significant communication or cognitive impairment on the part of the parent/caregiver that would preclude completion of questionnaires based on self-report.
2. the patient is a ward of the state or in foster care

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We expect to enroll 300 patients and one legal guardian per patient (parent or caregiver who has guardianship of the patient) per unit (for a total of 900 patients and 900 parents). A high-risk discharge assessment based on Mayo Clinic criteria will be used to identify children with complex or chronic conditions. Based on conversations with hospital leadership it is expected that approximately 120 patients per unit (40%) will have a complex or chronic condition. Parent experience related to quality of discharge teaching and care coordination will be self-reported by parents using established, reliable and valid scales. Child and parent characteristics, length of hospitalization, readmission, and Emergency Department use data will be extracted from electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Improved parent experience | 30 days
  Parents of children with and without complex or chronic health conditions who received enhanced discharge preparation by the clinical nurse using the SM-THINk protocol would report increased parent experience (quality of discharge teaching delivered and care coordination).

CONTACTS AND LOCATIONS:
Overall Officials: Stacee Lerret, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No